CLINICAL TRIAL: NCT07252037
Title: Impact of Dietary Guidelines Diets Containing Mostly Ultra-Processed Foods Compared to Less-Processed Foods on Biomarkers of Cardiometabolic Disease
Brief Title: Dietary Guidelines for Americans-Ultra Processed Study
Acronym: DGA-UP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Julie Hess, Research Nutritionist, USDA Grand Forks Human Nutrition Research Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: GFHNRC158
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Overweight , Obesity; Class I Obesity
Keywords: Healthy Weight; Stage I Hypertension
MeSH Terms: conditions — Overweight; Obesity; Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-processed DGA Diet (Experimental): Participants will be provided a Dietary Guidelines for Americans (DGA) compliant diet comprised of low-processed foods (Nova Categories 1-3)
  Interventions: Other: Low-processed DGA Diet
- Ultra-processed DGA Diet (Experimental): Participants will be provided a Dietary Guidelines for Americans (DGA) compliant diet comprised primarily of ultra-processed foods (Nova Category 4)
  Interventions: Other: Ultra-processed DGA Diet

INTERVENTIONS:
Other: Low-processed DGA Diet — Participants will consume a DGA menu made up of low-processed foods over a 4-week period
  Arms: Low-processed DGA Diet
Other: Ultra-processed DGA Diet — Participants will consume a DGA menu primarily made up of ultra-processed foods over a 4-week period
  Arms: Ultra-processed DGA Diet

SUMMARY:
The purpose of this research is to test how processing food can affect how one's body responds to it.

DETAILED DESCRIPTION:
The purpose of this project is to address the current gap in research on ultra-processed foods (UPFs) and cardiometabolic health with a feeding study that addresses the limitations of previously conducted intervention studies in matching UPF- and unprocessed- foods intervention diets for diet quality, nutrient content, and food type. Therefore, the primary objective is to evaluate diets composed primarily of ultra-processed or less processed foods that meet dietary guidelines recommendations on chronic disease risk factors. More specifically, when Dietary Guidelines for Americans (DGA)-compliant diets comprised of mostly ultra-processed and unprocessed foods (per Nova) are fed to generally healthy participants, determine whether there is an impact on:

* blood pressure
* fasting glucose and insulin concentrations, or
* lipid panel (total cholesterol, HDL-C, LDL-C, triglycerides).

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5-34.9 kg/m2
* Systolic <139 mm Hg and Diastolic <90 mm Hg
* Able to understand and sign the consent form
* Have own transportation to the Grand Forks Human Nutrition Research Center
* Not allergic to study foods or unwilling to eat them
* Willing to comply with study demands
* Able to read and understand English

Exclusion Criteria:

* Taking statins or medication to lower blood pressure,
* Taking anti-inflammatory or anti-diabetes medications
* Pregnant, lactating, or planning to become pregnant
* Diagnosed with an eating disorder
* Taking weight loss medications
* Smoke or use other tobacco products, including e-cigarettes
* Have overt hypothyroidism
* Diagnosed with cancer
* Exercise more than 30 minutes per day 2 or more days per week
* Allergic to study foods
* Express unwillingness to consume study foods at the screening appointment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Change in blood pressure from baseline | Week 0, Week 4

SECONDARY OUTCOMES:
Change in fasting and postprandial glucose and insulin concentrations from baseline | Week 0, Week 4
Change in lipid panel measures (total cholesterol, HDL-C, LDL-C, triglycerides) from baseline | Week 0, Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Julie Hess, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No